CLINICAL TRIAL: NCT04515732
Title: Prevalence, Pattern and Disease Course og Arthritis and Enthesitis in Patients With Psoriasis, and Effect of Apremilast in Subclinical, US-defined Psoriatic Arthritis - a Population Based Study Applying Clinical, Ultrasonic, MRI and Patient-reported Outcomes
Brief Title: Danish Population-based Assessment of Psoriasis and Psoriatic Arthritis (DANPAPP)
Acronym: DANPAPP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Professor Mikkel Østergaard (Other)
Collaborators: Celgene Corporation (Industry); The Danish Rheumatism Association (Other); The Danish Psoriasis Association (Unknown)
Responsible Party: Sponsor-Investigator, Professor Mikkel Østergaard, Professor, DMSc, PhD, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DANPAPP; 2016-004354-15 (EudraCT Number)
Record Dates: First submitted 2018-12-12; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Psoriasis; Psoriatic Arthritis
Keywords: Ultrasound; Patient reported outcome measures
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic | interventions — apremilast

STUDY DESIGN:
Intervention Model Description: As described. Only part 3 of the study is considered interventional.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3a (apremilast intervention) (Experimental): Apremilast in standard dosis (gradual increase 0-30 mg x 2 daily over the first 6 days, hereafter 30 mg x 2 daily) for 6 months, followed by 6 months observation.
  Interventions: Drug: Apremilast Oral Tablet
- 3b (non-intervention) (No Intervention): Observation

INTERVENTIONS:
Drug: Apremilast Oral Tablet — As in description
  Arms: 3a (apremilast intervention)

SUMMARY:
3-part study of patients with psoriasis, including 1) a population based questionnaire 2) cross-sectional clinical study with focus on musculoskeletal ultrasound and patient reported outcomes 3) 12 months follow-up study of patients with certain ultrasonic signs of psoriatic arthritis. Patients with pain: Interventional with 6 months treatment with apremilast, followed by 6 months observation. Patients without pain: 12 months observation.

DETAILED DESCRIPTION:
Part 1:

A population-based survey of Danish inhabitants, will by screening of approximately 10.000 Danes identify approximately 425 persons who report to have psoriasis(PsO) with or without psoriatic arthritis (PsA). These will receive an e-mail invitation to an internet based questionnaire regarding demographics, skin and joint complaints, diagnosed diseases, contact to health care providers, and different aspect of psychological and physical function and wellbeing (incl. function, health-related quality of life, depression, anxiety, social participation, and sleep disturbances). In the questionnaire the participant will be asked if he/she would be interested in participating in a clinical study.

Part 2:

Participants who accept the above mentioned invitation (estimated 273) will be seen in a Department of Rheumatology, for the following examination programme: Clinical examination with a focus on skin, joints and entheses,ultrasonic (US) examination of joints and entheses, patient-reported outcomes and blood sampling for both stratification and identification of biochemical signs of inflammation.

Patients with musculoskeletal pain and certain joint and/or entheseal inflammation documented by US, will be invited to participate in a 12 months' interventional study (part 3a, below), whereas patients without musculoskeletal pain but with US findings (as above) will be invited to participate in a 12 months non-interventional follow-up study (part 3b, below). Patients with pre-diagnosed PsA that by US have active inflammation (same definition and criteria as above), will also be invited to participate in the interventional study if they fit the criteria, especially those described under concomitant medication, otherwise they will be offered to participate in the non-interventional study.

Part 3a:

Patients with musculoskeletal pain in relation to joints and/or entheses (that is not explained by alternative diagnosis, as assessed by including rheumatologist) and "US-defined PsA", i.e. with certain joint and/or entheseal inflammation as documented by US, will be offered inclusion in a 12 months' interventional study, in which 6 month induction therapy with apremilast (in addition to their usual therapy) will be followed by cessation of apremilast and 6 months of observation. Patients will be followed with clinical examination, PRO's, blood sampling and US at months 3, 6, 9 and 12.

MRI will be performed at inclusion and at 6 months follow-up in selected patients (patients with dactylitis or with enthesitis in the ankle region (Achilles enthesitis or plantar fasciitis)).

Part 3b:

Patients without musculoskeletal pain but with certain joint or entheseal inflammation verified by US will be offered inclusion in a 12 months' non-interventional study. Patients will continue their current therapy and be followed with clinical examination, patient-reported outcomes, blood sampling and US at months 3, 6, 9 and 12.

ELIGIBILITY:
Inclusion Criteria:

In general (all parts of the study):

* Age >18 years
* Being able and willing to comply with the requirements of this protocol
* Having signed informed consent

Part 2:

• Psoriasis, diagnosed by a physician according to patient

Part 3a:

* Musculoskeletal pain in relation to joints or entheses (that is not explained by alternative diagnosis, as assessed by including rheumatologist) and"US-defined PsA" (ie. with certain joint and/or entheseal inflammation as documented by US (see 'Definitions of patient populations' for definition))
* MRI substudy:

  * Clinical dactylitis or enthesitis in the ankle region (Achilles enthesitis or plantar fasciitis)
  * No contraindications for MRI (see appendix 22.2.2) For allowed and disallowed previous and concomitant treatment, please see paragraph on "Previous and concomitant medication".

Part 3b:

• Not having musculoskeletal pain but still "US-defined PsA" (i.e. with certain joint and/or entheseal inflammation as documented by US (see 'Definitions of patient populations' for definition))

Exclusion Criteria:

In general (all parts of study):

• Incapability of complying with the examination program of this protocol for physical, mental or practical reasons.

Part 2:

• Incapability of understanding spoken or written danish.

Part 3a:

* Pregnancy, pregnancy wish or breast-feeding.
* Hypersensitivity to the active substance (apremilast) or any of the excipients.
* Hereditary problems of galactose intolerance, lactase deficiency or glucose-galactose
* malabsorption
* Severe renal failure (glomerular filtration rate (GFR) <30ml/min)
* Current treatment with potent CYP3A4 enzyme inhibitors (rifampicin, phenobarbital, carbamazepin, phenytoin, perikon ("grønne lykkepiller" , Neurokan, Modigen, Calmigen, Velzina))
* Current or planned (during the study period) treatment that might cause psychiatric symptoms
* Known active tuberculosis (TB) or history of incompletely treated TB.
* Clinical history of serious liver disease.
* Hepatitis B antigen positivity or Hepatitis C antibodies positivity at screening (tests ≤3 months before inclusion is accepted).
* Bacterial infections requiring antibiotics (oral or intravenously) or serious viral or fungal infections within the last four weeks before screening. Treatment of such infections should be completed 4 weeks prior to screening.
* Clinical history of serious immunological disease (including HIV or other congenital or acquired immune disease) or other serious uncontrolled disease.
* Current depression, previous depression, previous suicidal thoughts/tendencies or psychiatric symptoms
* Conditions, including abnormal laboratory measurements, which might put the patient at an unnecessary risk by participation in the study or make data difficult to interpret.
* Known inflammatory rheumatic disease other than PsA.
* MRI substudy: Contraindications for MRI (see appendix 22.2.2)
* Certain previous and concomitant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2018-12-14 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with PsO reporting musculoskeletal pain within the past 12 months | 1 day (At completion of questionnaire (performed once))
  Part 1 - e-based questionnaire. Number of patients reporting joint- or entheseal pain within the past 12 months
The difference in number of joints with US defined synovitis, in PsO patients with, compared to patients without musculoskeletal pain. | Day 0
  Part 2 - cross sectional study
The difference in number of entheses with US defined enthesitis, in PsO patients with, compared to patients without musculoskeletal pain. | Day 0
  Part 2 - cross sectional study
Change in OMERACT-EULAR Global US score of synovitis, from baseline to 6 months, in patients treated with apremilast (intervention group). | 6 months
  Part 3 - follow up study

SECONDARY OUTCOMES:
The correlations between presence of musculoskeletal pain and patient reported outcomes of function, health related quality of life, and impact on patient's lives (including EQ5D, HAQ and PsAID) | 1 day (At completion of e-based questionnaire (performed once))
  Part 1
The prevalence of US defined synovitis at the individual 48 joints sites in patients with compared to patients without musculoskeletal pain. | Day 0
  Part 2
The prevalence of US defined enthesitis at the individual 12 entheseal sites in patients with compared to patients without musculoskeletal pain. | Day 0
  Part 2
The correlation between clinical and US scores of synovitis and enthesitis with patient reported outcomes of pain, function and impact on patient's lives (including pain, HAQ and PsAID). | Day 0
  Part 2
Sensitivity and specificity of screening questionnaires, with fulfillment of CASPAR criteria as gold standard, and "US defined PsA" as alternative. | Day 0
  Part 2
Change in "US total count of inflamed joints and entheses" from baseline to 3, 6 and 12 months, and from 6 to 12 months, in intervention and non-intervention groups. | 3, 6, 12 months
  Part 3
Change in patient global pain on a visual analogue scale (VAS, range 0-100), from baseline to 6 months and from 6 to 12 months in intervention group. | 0-6 months, 6-12 months
  Part 3
Change in OMERACT-EULAR Global US score of synovitis from baseline to 3 and 6 months, and from 6 to 12 months, in intervention and non-intervention groups. | 0-3-6-12 months
  Part 3
Change in US enthesitis activity score from baseline to 3, 6 and 12 months, and from 6 to 12 months, in intervention and non-intervention groups. | 0-3-6-12 months
  Part 3
Change in PRO's (including PsAID, HAQ) from baseline to 3, 6, 9 and 12 months. | 0-3-6-9-12 months
  Part 3
The correlation between changes in clinical and US scores of synovitis and enthesitis and changes in patient reported outcomes, overall and in intervention and non-intervention groups. | 0-3-6-12 months
  Part 3

OTHER OUTCOMES:
Change in DAS28-CRP (Disease Activity Score, 28 joints, CRP) from baseline to month 3 and 6, and from month 6 to month 12. | 0-3-6-12 months
  Part 3
Change in PASDAS (Psoriatic Arthritis Disease Activity Score) from baseline to month 3 and 6, and from month 6 to month 12. | 0-3-6-12 months
  Part 3
Change in DAPSA (Disease Activity Index for Psoriatic Arthritis) from baseline to month 3 and 6, and from month 6 to month 12. | 0-3-6-12 months
  Part 3
Change in mCPDAI (modified Composite Psoriatic Disease Activity Index) from baseline to month 3 and 6, and from month 6 to month 12. | 0-3-6-12 months
  Part 3
Evaluation of EULAR response criteria from baseline to month 3 and 6, and from month 6 to month 12. | 0-3-6-12 months
  Part 3
Evaluation of ACR (American College of Rheumatology) response criteria from baseline to month 3 and 6, and from month 6 to month 12. | 0-3-6-12 months
  Part 3
Evaluation of PsARC (Psoriatic Arthritis Response Criteria) from baseline to month 3 and 6, and from month 6 to month 12. | 0-3-6-12 months
  Part 3

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Videncenter for Reumatologi og Rygsygdomme, Rigshospitalet Glostrup, Glostrup Municipality
  - Dansk Gigthospital, Sønderborg